CLINICAL TRIAL: NCT03490747
Title: Clinical and Cost-effectiveness of a Co-developed, Evidence-based Physical Activity Referral Scheme for the Treatment and Prevention of Health Conditions: a Pragmatic Trial
Brief Title: Evaluation of a Physical Activity Referral Scheme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paula Watson (Other)
Collaborators: University of Bath (Other); University of Gloucestershire (Other); University of Liverpool (Other); Brock University (Other); Radboud University Medical Center (Other)
Responsible Party: Sponsor-Investigator, Paula Watson, Senior Lecturer, Liverpool John Moores University
Organization: Liverpool John Moores University (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: SPS-17-01
Record Dates: First submitted 2018-01-11; First posted 2018-04-06 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Cardiovascular Risk Factor; Diabetes Mellitus, Type 2; Anxiety; Depression; Musculoskeletal Injury; Cardiovascular Diseases; Cancer; Obesity; Metabolic Syndrome; Physical Activity
Keywords: Physical Activity; Pragmatic Evaluation; Exercise Referral; Mixed-methods; Behaviour Change; Intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Anxiety Disorders; Depression; Cardiovascular Diseases; Neoplasms; Obesity; Metabolic Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: 3 arm quasi-experimental trial
  1. Co-developed scheme 2. Usual care 3. No treatment control
Who Masked: Outcomes Assessor
Masking Description: Post hoc data analysis will be blinded via an independent coding method for condition and time frame (i.e. pre-post measures).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Co-developed referral scheme (Experimental): A physical activity referral scheme co-developed by multidisciplinary stakeholders to incorporate behaviour change support and ensure pragmatic relevance and feasibility.
  Interventions: Behavioral: Physical activity referral scheme
- Usual care referral scheme (Active Comparator): Comparative, usual care exercise referral scheme.
  Interventions: Behavioral: Usual care exercise referral scheme
- No treatment control (No Intervention): Lifestyle advice leaflet only (provided to participants in all arms during baseline assessments).

INTERVENTIONS:
Behavioral: Physical activity referral scheme — An 18-week physical activity referral scheme co-developed by a local multidisciplinary stakeholder group. Behaviour change support underpinned by Self-Determination Theory (Ryan & Deci, 2000) will be provided by an exercise referral practitioner at weeks 1,4,8,12 and 18 to facilitate increased physical activity levels. Patients will be supported to develop a tailored programme of physical activity that may involve use of the fitness centre facilities (e.g. swimming, group classes, gymnasium use), participation in community-based initiatives, and changes to habitual physical activity. Focus on promoting patient autonomy and tailoring activities to patient's preferences and needs. Subsidised access to fitness centre facilities for first 12 weeks.
  Arms: Co-developed referral scheme
Behavioral: Usual care exercise referral scheme — A comparative usual care exercise referral scheme that includes fitness centre based activities (e.g. swimming, group classes, gymnasium use). Patients meet an exercise referral practitioner at their induction (week 1) and week 12 (post scheme). Patients are typically prescribed a gym-based, 12-week programme. Subsidised access to fitness centre facilities for 12 weeks.
  Arms: Usual care referral scheme

SUMMARY:
The study will evaluate the effectiveness of a co-developed exercise referral scheme. Participants will be recruited to one of three groups 1. Co-developed exercise referral scheme, 2. Usual care exercise referral scheme, 3. No treatment control (no intervention). The study will measure effectiveness by observing change in cardiorespiratory fitness at 12 weeks. Intervention cost-effectiveness will also be evaluated at 3 months follow-up using objective physical activity data.

DETAILED DESCRIPTION:
Evidence of effectiveness for UK exercise referral is unclear. This representation has been deemed an unfair assessment of its potential to impact public health. This is due to systematic review evidence that reports evaluations of exercise referral interventions that are not evidence-based or underpinned by behaviour change theory.

This evaluation is the third phase of a project that aims to co-develop (Phase 1), pilot (phase 2) and evaluate (phase 3) an evidence-based exercise referral scheme. This approach is underpinned by the Medical Research Council guidance for complex interventions.

Through co-development work with a multidisciplinary group of researchers and local stakeholders and subsequent pilot work, it is hypothesised that the co-developed, evidence-based intervention will have improved chances of implementation success, and therefore, clinical effectiveness.

ELIGIBILITY:
Inclusion Criteria:

• 18 years or older and have a health-related risk factor (e.g. high blood pressure, hyperglycaemia, obesity etc.) or a health condition (diabetes, cardiovascular disease, anxiety, depression etc.) that may be alleviated by increasing current PA levels.

Exclusion Criteria:

* Uncontrolled health-conditions (Cardiac, metabolic, respiratory etc.) and/or any recent traumatic events (e.g. myocardial infarction).
* Unstable angina or aortic stenosis.
* Severe psychological or neurological conditions.
* Participation in an ERS at any location other than the research centres (at the time of recruitment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Change in cardiorespiratory fitness | Baseline and week 12.
  Estimated via the Astrand-Rhyming cycle protocol using the updated age and sex specific nomogram.

SECONDARY OUTCOMES:
Change in objective physical activity levels | Baseline, week 12, and 6 months
  Objective physical activity levels will be analysed using a hip worn accelerometer (ActiGraph GT3X). 7-day monitoring periods will recorded at three time points. During the 7-day monitoring period, each participant will complete a diary to record hours of use and to distinguish between work and leisure hours.
Change in flow-mediated dilation | Baseline and week 12.
  Endothelium dependent vasodilatation of the brachial arteries will be examined using ultrasound. Brachial artery baseline diameter and blood flow will be assessed in one arm. An ultrasound probe is placed on the bicep for 1 minute before a blood pressure cuff (placed around the forearm) is inflated to suprasystolic pressure (~220 mmHg) for 5 minutes. Immediately after the cuff is deflated, changes in arterial diameter and flow will be assessed continuously for 3 minutes using the ultrasound probe. Ultrasound data will then be analysed post hoc.
Change in carotid vasoreactivity | Baseline and week 12.
  The carotid vasoreactivity (cold pressor) test will measure the carotid artery's response to a stimulus. Similar to the flow-mediated dilation procedure, an ultrasound probe will be placed on the patient's left side of their neck, positioned in such a way to allow a clear image of the right common carotid artery to be displayed on the ultrasound monitor screen. The cold pressor procedure involves submersion of the left hand to wrist in ice slush for 180-seconds. Ultrasound data will then be analysed post hoc.
Change in total cholesterol | Baseline and week 12.
  A 15ml blood sample will be taken. Blood profiles will be analysed as a measure of cardiometabolic health. Analysis will be conducted at LJMU. Patients will be made aware of the storage and use of their tissue.
Change in plasma glucose | Baseline and week 12.
  A 15ml blood sample will be taken. Blood profiles will be analysed as a measure of cardiometabolic health. Analysis will be conducted at LJMU. Patients will be made aware of the storage and use of their tissue.
Change in triglycerides | Baseline and week 12.
  A 15ml blood sample will be taken. Blood profiles will be analysed as a measure of cardiometabolic health. Analysis will be conducted at LJMU. Patients will be made aware of the storage and use of their tissue.
Change in self-reported physical activity | Baseline, week 12, and 6 months.
  Patients' perceived physical activity levels will be recorded with the short version of the International Physical Activity Questionnaire (IPAQ, Craig et al., 2003). The short-IPAQ is a 7-day recall self-administered tool that measures intensity, frequency and duration of physical activity and provides a total estimate of energy expenditure. A total score of MET-minutes/day/week and sedentary behaviour minutes/day/week will be calculated according to the IPAQ scoring protocol.
Change in psychological wellbeing | Baseline, week 12, and 6 months.
  Psychological wellbeing will be measured using the Warwick-Edinburgh Mental Well-being Scale (WEMWBS, Tennant et al., 2007). WEMWBS is a 14-item positively worded instrument containing items related to psychological functioning (e.g. "I've been thinking clearly") and subjective well-being (e.g. "I've been feeling cheerful"). Participants are asked to rate on a Likert scale of 1 (none of the time) to 5 (all of the time) how well each statement describes their experiences over the last two weeks.
Attendance at consultations | Week 1, 4, 8, 12, and 18
  Patient attendance records will be collected by ERPs at the following time-points:
  * Intervention centre: 1, 4,8,12 and 18 weeks;
  * Usual care centre: 1 and 12 weeks.
Attendance at fitness centre | Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12. Months 4, 5 and 6
  The number of times patients sign in at the fitness centre to go to either the gym or a class will be recorded on a weekly basis for weeks 1 to 12, then on a monthly basis up to 6 months. This information is automatically recorded at fitness centres when patients visit.
Fidelity - consultation attendance | Week 18
  ERPs from both intervention and usual care centres will be asked to monitor the number of consultations offered (measured by appointment bookings or records of appointments offered but declined by participants), and the number of consultations conducted for each patient.
Fidelity - consultation communication strategies | Week 1, 4, 8, 12, and 18
  A random sample of ERS inductions from both intervention and usual care centres (approx 10 per centre) plus a random sample of 4, 8, 12 and 18-week consultations from the intervention centre only will be audio-recorded and coded for the use of "needs-supportive" communication strategies (using a coding manual developed through a previous pilot study (REF 16/WA/0231)). In addition, all intervention centre recordings will be coded for fidelity to an agreed protocol, e.g. asking required questions about physical activity, setting an action plan, giving out patient log book etc.
Change in health-related quality of life measure | Baseline, week 12, and 6 months.
  Participants' change in health-related quality of life (HRQoL) will be measured at baseline, 12 weeks, and 6 months. The EQ-5D will be used, this is a validated tool for measuring HRQoL. This tool has been applied successfully in a recent UK trial-based economic evaluation of exercise referral schemes (Edwards et al. 2013).
Intervention operating and set up costs | Week 18
  Captured via telephone interview with Exercise Referral Scheme Personnel from (organisation e.g. local authority/ fitness centre/ research institute; questions adapted from validated questionnaire).
Loss in revenue costs | Week 18
  Captured via telephone interview with fitness centre manager and/or coordinators (questions have been used in previous research).
Change in patient costs | Baseline, Week 12 and 6 months
  Captured via patient questionnaire during lab testing (questions adapted from validated questionnaire).
Change in patient health care utilisation costs | Baseline and 6 months
  Captured via questionnaire (questions adapted from validated questionnaire).

OTHER OUTCOMES:
Change in exercise motivation | Baseline, week 12, and 6 months.
  The Behavioural Regulation in Exercise Questionnaire (BREQ-2, Markland & Tobin, 2004) plus 4 additional items (Wilson et al., 2006a) will be used to assess exercise motivation. The BREQ-2 is a widely-used instrument comprised of 19 items describing reasons why people exercise (e.g. "I think exercising is a waste of time"; "I feel ashamed when I miss an exercise session"; "I exercise because it's fun"). Participants answer on a likert scale of 0 (not true for me) to 4 (very true to me) to indicate how true each item is for them.
Change in psychological needs satisfaction | Baseline, week 12, and 6 months.
  Psychological need satisfaction will be measured using the Psychological Need Satisfaction in Exercise Scale (PNSE, Wilson et al., 2006b). The PNSE is an 18-item instrument designed to measure participants' perceived autonomy (e.g. "I feel free to exercise in my own way"), competence (e.g. "I feel capable of completing exercises that are challenging to me") and relatedness (e.g. "I feel connected to the people who I interact with while we exercise together") in an exercise context. Participants are asked to answer on a 6-point likert scale (1 = false, 6 = true) to indicate how they typically feel when they exercise.
Change in perceived needs support | Baseline, week 12, and 6 months.
  Needs support will be measured using a 15-item needs support (NS) tool developed by Markland and Tobin (2010) to measure the extent to which participants perceive their exercise instructors provide support for autonomy, structure (linked to competence) and involvement (linked to relatedness).
Change in intentions to engage in physical activity | Baseline, week 12, and 6 months.
  Three items developed by Edmunds et al. (2007) will be used to assess patients' intentions to engage in PA (e.g. "I plan to regularly engage in PA during the next 3 months").
Patient focus groups - intervention | Week 12
  Focus groups will be conducted with a purposeful subsample of patients after approximately 6-12 weeks of attending the scheme (e.g. those with low attendance, high attendance, significant health changes, no change etc.). Two focus groups will be conducted with patients attending the intervention centre (approx 5-8 participants per group). Focus groups will be conducted at the individual fitness centres and will last approximately 60 minutes. Discussion will focus on the extent to which, and how, patients feel each ERS is facilitative (or not) in helping them become more physically active, with questions about staff interactions, activities on offer, and the impact of the scheme on their likely continuation with physical activity.
Patient focus groups - usual care | Week 12
  Focus groups will be conducted with a purposeful subsample of patients after approximately 6-12 weeks of attending the scheme (e.g. those with low attendance, high attendance, significant health changes, no change etc.). Two focus groups will be conducted with patients attending the usual care centre (approx 5-8 participants per group). Focus groups will be conducted at the individual fitness centres and will last approximately 60 minutes. Discussion will focus on the extent to which, and how, patients feel each ERS is facilitative (or not) in helping them become more physically active, with questions about staff interactions, activities on offer, and the impact of the scheme on their likely continuation with physical activity.
Exercise referral practitioner (ERP) interviews (intervention group only) | Week 18
  ERPs from the intervention centre only will take part in a semi-structured interview (after over half of patients have reached the 18-week point). The interviews will aim to explore the acceptability of the co-developed intervention, any challenges of delivery, and areas that require further development etc.

CONTACTS AND LOCATIONS:
Overall Officials: Paula M Watson, PhD, Principal Investigator — Liverpool John Moores University
Locations (1):
- Liverpool John Moores University, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buckley BJ, Thijssen DH, Murphy RC, Graves LE, Cochrane M, Gillison F, Crone D, Wilson PM, Whyte G, Watson PM. Pragmatic evaluation of a coproduced physical activity referral scheme: a UK quasi-experimental study. BMJ Open. 2020 Oct 1;10(10):e034580. doi: 10.1136/bmjopen-2019-034580. PMID 33004383

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/47/NCT03490747/Prot_SAP_001.pdf